CLINICAL TRIAL: NCT07159880
Title: Extended Therapy Versus Traditional Therapy With Letrozole for Ovulation Induction in Women With Polycystic Ovary Syndrome: A Randomized Controlled Trial
Brief Title: Letrozole Extended vs Traditional Therapy for Ovulation Induction in Women With PCOS (PROLEx-PCOS)
Acronym: PROLEx-PCOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GABRIEL MONTEIRO PINHEIRO (Other)
Responsible Party: Sponsor-Investigator, GABRIEL MONTEIRO PINHEIRO, Study Director, Obstetrician and Gynecologist, Department of Obstetrics and Gynecology, Hospital Wladimir Arruda; Professor of Obstetrics and Gynecology, University of Santo Amaro (UNISA), EMBRIONARE
Organization: EMBRIONARE (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 88592925.0.0000.0081
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: PCOS (Polycystic Ovary Syndrome); Infertility; Anovulation
Keywords: polycystic ovary syndrome; PCOS; Ovulation induction; Letrozole; Aromatase Inhibitor; Extended letrozole therapy; traditional letrozole therapy; standart letrozole therapy; infertility; anovulation; ovulation rate; pregnancy rate
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility; Anovulation

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, parallel assignment clinical trial designed to compare extended letrozole therapy with standard letrozole therapy for ovulation induction in women with polycystic ovary syndrome (PCOS). Participants will be randomized in a 1:1 ratio into two groups: extended therapy (letrozole 5 mg/day from cycle days 2-12) and standard therapy (letrozole 5 mg/day from cycle days 2-6). Ovulation will be monitored by transvaginal ultrasound and confirmed with urinary LH testing. The primary outcome is ovulation rate. Secondary outcomes include number and size of mature follicles, clinical pregnancy rate, miscarriage rate, multiple pregnancy rate, time to conception, and incidence of ovarian hyperstimulation syndrome (OHSS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Letrozole Therapy (Active Comparator): Participants in this group will receive standard letrozole therapy for ovulation induction. Letrozole will be administered orally at a dose of 5 mg/day from cycle day 2 through cycle day 6 (5 consecutive days). Ovulation monitoring will be performed by transvaginal ultrasound and confirmed with urinary LH testing and/or corpus luteum visualization. This arm serves as the active comparator against the extended regimen for evaluating efficacy and safety outcomes.
  Interventions: Drug: Traditional Letrozole Therapy
- Extended Letrozole Therapy (Experimental): Participants in this group will receive extended letrozole therapy for ovulation induction. Letrozole will be administered orally at a dose of 5 mg/day from cycle day 2 through cycle day 12 (10 consecutive days). Ovulation monitoring will be performed by transvaginal ultrasound and confirmed with urinary LH testing and/or corpus luteum visualization. This arm will be compared with the standard regimen to assess differences in ovulation rate, follicular development, pregnancy outcomes, and safety.
  Interventions: Drug: Extended Letrozole Therapy

INTERVENTIONS:
Drug: Traditional Letrozole Therapy — Traditional therapy group: 5 mg/day of letrozole for 5 days (cycle days 2-6).
  Arms: Traditional Letrozole Therapy
Drug: Extended Letrozole Therapy — Extended therapy group: 5 mg/day of letrozole for 10 days (cycle days 2-12)
  Arms: Extended Letrozole Therapy

SUMMARY:
This randomized clinical trial aims to compare the efficacy and safety of extended letrozole therapy (5 mg/day for 10 days) versus standard letrozole therapy (5 mg/day for 5 days) for ovulation induction in women with polycystic ovary syndrome (PCOS). A total of 84 women aged 18-40 years will be randomized into two groups. Ovulation will be monitored by transvaginal ultrasound and confirmed with urinary LH testing and/or corpus luteum presence. The primary outcome is ovulation rate, while secondary outcomes include number and size of mature follicles, clinical pregnancy rate, multiple pregnancy rate, miscarriage rate, number of cycles until pregnancy, and incidence of ovarian hyperstimulation syndrome (OHSS).

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a prevalent endocrine disorder and one of the leading causes of anovulatory infertility worldwide. Letrozole, an aromatase inhibitor, has emerged as the preferred first-line pharmacological agent for ovulation induction in women with PCOS. Despite its widespread use, there is ongoing debate regarding the optimal duration of therapy to maximize ovulatory and pregnancy outcomes.

This randomized clinical trial is designed to evaluate whether an extended regimen of letrozole provides superior reproductive outcomes compared with the standard regimen. The extended protocol consists of daily administration of 5 mg letrozole from cycle day 2 through day 12, whereas the standard regimen involves 5 mg daily from cycle day 2 through day 6. Ovulatory response will be monitored through serial transvaginal ultrasound and biochemical markers of ovulation.

The trial aims to generate high-quality evidence on the efficacy and safety of extended letrozole therapy. The findings may inform future clinical guidelines on ovulation induction strategies in women with PCOS and contribute to optimizing treatment protocols for anovulatory infertility.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 40 years;
* BMI between 18,5 and 31 kg/m2
* Diagnosis of Polycystic Ovary Syndrome (PCOS) according to the Rotterdam criteria (2003) (presence of at least two of the following: oligo/anovulation, clinical and/or biochemical hyperandrogenism, polycystic ovarian morphology on ultrasound);
* Active desire for pregnancy at the time of enrollment;
* Ability and willingness to provide written informed consent (ICF).

Exclusion Criteria:

* Age <18 or >40 years;
* Presence of confirmed bilateral tubal factor, severe male factor infertility, premature ovarian insufficiency, uncontrolled hyperprolactinemia or thyroid dysfunction);
* Congenital or acquired uterine malformations;
* History of gynecologic or breast cancer;
* Known hypersensitivity to, or contraindication for, letrozole;
* Severe uncontrolled systemic disease (e.g., cardiovascular, renal, or hepatic disorders);
* Pregnancy or breastfeeding at the time of screening.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Ovulation rate | Assessed within one treatment cycle (up to 6 weeks from the start of medication).
  Proportion of participants achieving ovulation, defined as the presence of a dominant follicle ≥18 mm on transvaginal ultrasound with confirmation by urinary LH surge and/or visualization of corpus luteum.

SECONDARY OUTCOMES:
Clinical Pregnancy Rate | Assessed within 8 weeks after the start of treatment.
  Proportion of participants achieving clinical pregnancy, defined as visualization of a gestational sac by transvaginal ultrasound.
Number of Mature Follicles | Assessed during one treatment cycle (up to 6 weeks).
  Number of follicles ≥18 mm observed by transvaginal ultrasound in the stimulated cycle.
Follicular Size | Assessed during one treatment cycle (up to 6 weeks).
  Maximum diameter (in millimeters) of the leading follicle(s) observed by transvaginal ultrasound.
Miscarriage Rate | Assessed up to 12 weeks of gestation.
  Proportion of participants with spontaneous pregnancy loss within the first trimester (<12 weeks of gestation).
Multiple Pregnancy Rate | Assessed within 8 weeks after the start of treatment.
  Proportion of participants with multiple gestations, confirmed by transvaginal ultrasound.
Incidence of Ovarian Hyperstimulation Syndrome (OHSS) | Assessed within one treatment cycle (up to 6 weeks).
  Proportion of participants presenting clinical or ultrasound signs of OHSS during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel M Pinheiro, MD, Study Director — University of Santo Amaro; Katherine Ann R Miller, Medical student, Principal Investigator — Universisty of Santo Amaro
Locations (1):
- Health Complex Dr Wladimir Arruda, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be shared with qualified researchers with academic interest in polycystic ovary syndrome (PCOS), ovulation induction, or related reproductive medicine topics. Any shared data will be de-identified and coded, with no personal health information (PHI) included. Approval of the request by the principal investigator and execution of all applicable agreements (e.g., data use agreement or material transfer agreement) will be required prior to data sharing.
Supporting Information: ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided only in accordance with participants' informed consent (ICF). For more information or to submit a request, please contact katherinereimao000@gmail.com